CLINICAL TRIAL: NCT03870412
Title: Multi-center, Open, One-arm Clinical Study Evaluating the Efficacy and Safety of Pegylated Recombinant Human Granulocyte-stimulating Factor Injection (PEG-rhG-CSF) in Preventing Neutropenia in Elderly Patients With Lymphoma After Chemotherapy
Brief Title: Evaluation of the Application of PEGylated Recombinant Human Granulocyte Stimulating Factor Injection (PEG-rhG-CSF) in Chemotherapy of Elderly Lymphoma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC Baike (Shandong) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CSPC-JYL-LY-03
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-02

CONDITIONS: Elderly Lymphoma Patients
Keywords: PEG-rhG-CSF
MeSH Terms: interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEG-rhG-CSF (Experimental): Jin Youli(PEG-rhG-CSF):From the first cycle of chemotherapy, Jin Youli(PEG-rhG-CSF) was injected subcutaneously 24-72 hours after the end of chemotherapy, 6 mg was given to patients with body weight ≥45 kg, and 3 mg was given for body weight <45 kg. Inject once every chemotherapy cycle.
  Interventions: Drug: PEG-rhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF — The test drug PEG-rhG-CSF was administered prophylactically to elderly lymphoma patients who met the inclusion/exclusion criteria 24-72 hours after chemotherapy.

SUMMARY:
A multicenter, open, one-arm clinical study evaluated the efficacy and safety of Jinyouli in preventing neutropenia after chemotherapy in elderly lymphoma patients who met the criteria for admission. Chemotherapy regimen: The investigator selected according to the specific condition the corresponding standard chemotherapy regimen, the chemotherapy regimen used, FN risk ≥ 20%, or 10% < FN risk < 20% with at least one high risk factor for FN, from the first cycle of chemotherapy, 24-72 after chemotherapy hour subcutaneous injection of Jinyouli.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥ 65 years, gender is not limited;
* (2) Patients with lymphoma diagnosed by histopathology or cytology;
* (3) Patients requiring multi-cycle chemotherapy;
* (4) Planned chemotherapy regimen FN risk ≥ 20 % (see Annex I), or 10% <FN risk < 20% (see Annex II) with high risk factors for at least one FN;
* (5) Physical status (KPS) score ≥ 70 points;
* (6) Expected Survival period of more than 3 months;
* (7) normal bone marrow hematopoietic function (ANC ≥1.5×109/L, PLT≥100×109/L, Hb≥80g/L, WBC≥3.0×109/L);
* (8) The testers (or their legal representatives/guardians) must sign an informed consent form.

Exclusion Criteria:

* (1) Lymphoma central involvement;
* (2) Hematopoietic stem cell transplantation or organ transplantation;
* (3) Insufficient local or systemic infection;
* (4) Severe internal organ dysfunction and occurred in the last 6 months Myocardial infarction;
* (5) Liver function tests total bilirubin (TBIL), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) are >2.5 times the upper limit of normal, if the above indicators are >5 times due to liver metastasis Upper limit of normal value; renal function test: serum creatinine (Cr) > 2 times the upper limit of normal;
* (6) allergic to PEG-rhG-CSF, rhG-CSF and other preparations or proteins expressed by Escherichia coli;
* (7) Severe mental illness, affecting informed consent and/or adverse reaction expression or observation;
* (8) The investigator judges patients who are not suitable for participation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 485 (Estimated)
Dates: Start 2019-02-22 (Actual); Primary Completion 2021-03-22 (Estimated); Study Completion 2021-08-22 (Estimated)

PRIMARY OUTCOMES:
Incidence of febrile neutropenia in cycles 1 to 6 | through 1-6 cycles of PEG-rhG-CSF,an average of 6 month
  The body temperature standard for neutropenic fever is sputum temperature; febrile neutropenia is defined as ANC < 0.5*109 / L and sputum temperature> 38.0 ° C.

SECONDARY OUTCOMES:
The incidence of grade IV neutropenia in the first to sixth cycles of PEG-rhG-CSF. | through 1-6 cycles of PEG-rhG-CSF,an average of 6 month
  The incidence of grade IV neutropenia in the first to sixth cycles of PEG-rhG-CSF.
Incidence of dose adjustment of chemotherapy drugs in each chemotherapy cycle | through 1-6 cycles of PEG-rhG-CSF,an average of 6 month
  Incidence of dose adjustment of chemotherapy drugs in each chemotherapy cycle
Incidence of chemotherapy delays in each chemotherapy cycle | through 1-6 cycles of PEG-rhG-CSF,an average of 6 month
  Incidence of chemotherapy delays in each chemotherapy cycle
The proportion of patients receiving antibiotics during the entire chemotherapy period. | through 1-6 cycles of PEG-rhG-CSF,an average of 6 month
  The proportion of patients receiving antibiotics during the entire chemotherapy period.

CONTACTS AND LOCATIONS:
Overall Officials: Huiqiang Huang, Principal Investigator — Sun Yat-sen University Cancer Hospital
Locations (1):
- Sun Yat-sen University Cancer Hospital, Guangzhou, China